CLINICAL TRIAL: NCT04644978
Title: European Study on the Attitude of Psychiatrists Towards Their Patients
Acronym: Eustigma
Status: Completed | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dorottya Ori, Principal investigator, MD, Semmelweis University
Other Study IDs: Eustigma - v. 1.0
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Mental Illness; Stigmatization
Keywords: Stigma; Mental health related stigma; Stigmatising attitude; Mental health problems; Survey; Psychiatry; Psychiatrist
MeSH Terms: conditions — Mental Disorders; Stereotyping; Social Stigma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trainees and specialists in child and adult psychiatry: The responder must be a practising specialist or trainee in psychiatry or child and adolescent psychiatry in the participating European countries on the basis of his / her own declaration. Responders could provide their consent by choosing "I agree" on the website, after reading the information leaflet and the informed consent form.
  Interventions: Other: anonymous online survey

INTERVENTIONS:
Other: anonymous online survey — An online questionnaire will be provided for the participants of our study. Participation in the study is voluntary and it can be terminated at any time without having to give any reasons.

SUMMARY:
Background: Many people think that people with mental disorders might be dangerous or unpredictable. These patients face various sources of disadvantages and experience discrimination on job interviews, in education, and housing. Mental health-related stigma (MHS) occurs not only within the public community, it is a growing issue among professionals as well.

Aim: The investigators designed a prospective, observational, multi-centre, international study of 35 European countries to investigate the MHS among medical specialists and trainees in the field of general adult and child and adolescent psychiatry.

Methods: An internet-based, anonymous survey will measure the stigmatizing attitude by using the local version of the Opening Minds Stigma Scale for Health Care Providers.

Presentation of the Results: The results of the research will be published in an international peer-reviewed journal. Furthermore, the research team will present the results at national and international conferences.

DETAILED DESCRIPTION:
There is a rising interest in the examination of the MHS that has been mostly studied among community people. Numerous international studies have shown that people with mental illness are considered to be unpredictable and dangerous. These people often experience disadvantages in various situations, like job interviews, education, and housing.

The MHS has been much less examined among medical professionals and psychiatrists; however, studies have shown that it is prevalent among them as well.

A recent multi-centre study collected the positive and negative experiences of 777 people with schizophrenia regarding access to healthcare services in 27 countries. More than 17% of the patients experienced some kind of discrimination due to their mental illness when they sought medical care for physical problems. More than 38% felt that the medical staff was disrespectful during psychiatric services. Higher discrimination was found within the former Eastern Bloc countries.

Generally, psychiatrists tend to be more empathetic towards people with mental illnesses; however, the MHS could be observed among them as well. A few studies have also shown that their attitude is more negative than that of community people.

Based on the ambiguous results and the lack of studies focusing on the stigmatizing attitude of psychiatrists, the research team aimed to examine this important issue among medical professionals in the mental health field.

Aim of the study:

Our aim is to investigate the stigmatizing attitudes and behaviours of adult psychiatric and child and adolescent psychiatric professionals and trainees towards people with mental illness in European countries.

The results of our study will contribute to the expansion of the existing knowledge both on national and international levels. The outcome could be used for the development of anti-stigma programs and the improvement of therapeutic options in the future.

Structure of the research:

Our study is cross-sectional and multi-centred across 35 European countries. The research team would like to measure the extent of the stigmatizing attitude and its relationship with psychosocial factors.

* Sociodemographic measures:

  * sociodemographic data: age, sex
  * professional data: workplace categories (university, psychiatric hospital, outpatient service, research centre); location of the workplace (capital, county seat, rural town, small town, village); years of professional experience; current psychotherapeutic activity
  * personal information (related to a stigmatizing attitude): mental illness is known in his/her family or close friend, previous treatment for own mental illness, attending psychotherapy
* National version of the Opening Minds Stigma Scale for Health Care Providers (OMS-HC)

An online questionnaire will be provided for the participants of our study. Participation in the study is voluntary, and it can be terminated at any time without having to give any reasons.

ELIGIBILITY:
Inclusion Criteria:

* The responder must be a practising specialist or trainee in psychiatry or child and adolescent psychiatry in one of the participating countries on the basis of his / her own declaration.
* Responders could provide their consent by choosing "I agree" on the website, after reading the information leaflet and the informed consent form. Only those participants will be able to complete the online survey who chose "I agree" on the website.

Exclusion Criteria:

* The choice of "I do not agree" option of the participant on the website after reading the informed consent form. The responder will be guided automatically to the end of the survey.

Min Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Practising specialists and trainees in adult psychiatry or child and adolescent psychiatry who work in the participating European countries
Sampling Method: Non-Probability Sample
Enrollment: 4245 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
stigmatising attitude | Baseline
  The main questionnaire is the Opening Minds Stigma Scale for Health Care Providers (OMS-HC) which is a self-report questionnaire that contains 15 statements describing feelings and opinions about people with mental health problems. . In the survey, the subjects indicate on a 5-point Likert scale (1 = "strongly disagree" to 5 = "strongly agree") the extent they identify themselves with the given statement.
  The overall stigmatising attitude of the participants is described with the total score of the scale (minimum of 15, and a maximum of 75 points). Besides the total score, three dimensions can be calculated by evaluating the three subscales of the questionnaire (Attitude, Disclosure and Help-seeking, and Social Distance).
  Higher scores on a subscale and higher total scores reflect a more stigmatising attitude.

CONTACTS AND LOCATIONS:
Overall Officials: Dorottya Ori, MD, Principal Investigator — Vadaskert Child and Adolescent Psychiatric Hospital, Budapest, Hungary
Locations (31):
- Xhavit Gjata Hospital, Tirana, Albania
- Department of Psychiatry and Psychotherapeutic Medicin, Medical University of Graz, Graz, Austria
- City Hospital N15, Baku, Azerbaijan
- Psychiatric Clinic of Minsk City, Minsk, Belarus
- Military Medical Academy, Department of Psychiatry, Sofia, Bulgaria
- University Hospital Centre Zagreb, Zagreb, Croatia
- Private Practice, Nicosia, Cyprus
- 3rd Faculty of Medicine, Charles University, Prague, Czechia
- Research Unit for Child and Adolescent Psychiatry, Psychiatry- Aalborg University Hospital, Aalborg, Denmark
- University of Tartu, Tartu, Estonia
- EPSM Étienne Gourmelen, Quimper, France
- Klinikum rechts der Isar der Technischen Universität München, Munich, Germany
- Department of Psychiatry, Faculty of Medicine, School of Health Sciences, University of Ioannina, Ioannina, Greece
- Semmelweis University, Budapest, Hungary
- Department of Liasion Psychiatry, Mater University Hospital, Dublin, Ireland
- University Magna Graecia of Catanzaro, Catanzaro, Italy
- Hospital Gintermuiza, Jelgava, Latvia
- Vilnius University, Facutly of Medicine, Psychiatric Clinic, Vilnius, Lithuania
- Mount Carmel Hospital, Attard, Malta
- Clinical Centre of Montenegro, Clinic for Psychiatry, Podgorica, Montenegro
- Erasmus University, Rotterdam, Netherlands
- Institute of Psychological Medicine, Faculty of Medicine of University of Coimbra, Coimbra, Portugal
- The Serbsky State Scientific Center for Social and Forensic Psychiatry, Moscow, Russia
- Institute for Mental Health, Belgrade, Serbia
- Psychiatric Hospital Michalovce, Michalovce, Slovakia
- Centre for Clinical Psychiatry, University Psychiatric Clinic and Children's hospital Ljubljana, Ljubljana, Slovenia
- Fidmag Foundation, Barcelona, Spain
- Psychiatrische Klinik Clienia Littenheid, Littenheid, Switzerland
- Ankara City Hospital Bilkent, Ankara, Turkey (Türkiye)
- Chernivtsi Regional Mental Hospital, Bukovinian State Medical University, Chernivtsi, Ukraine
- Pennine Care NHS Foundation Trust, Oldham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ori D, Szocsics P, Molnar T, Motlova LB, Kazakova O, Morkl S, Wallies M, Abdulhakim M, Boivin S, Bruna K, Cabacos C, Carbone EA, Dashi E, Grech G, Greguras S, Ivanovic I, Guevara K, Kakar S, Kotsis K, Ingeholm Klinkby IM, Maslak J, Matheiken S, Mirkovic A, Nechepurenko N, Panayi A, Pereira AT, Pomarol-Clotet E, Raaj S, Prelog PR, Soler-Vidal J, Strumila R, Schuster F, Kisand H, Reim A, Ahmadova G, Vircik M, Kafali HY, Grinko N, Gyorffy Z, Rozsa S. Attitudes of psychiatrists towards people with mental illness: a cross-sectional, multicentre study of stigma in 32 European countries. EClinicalMedicine. 2023 Dec 6;66:102342. doi: 10.1016/j.eclinm.2023.102342. eCollection 2023 Dec. PMID 38149261